CLINICAL TRIAL: NCT01426087
Title: Investigator Sponsored Study of Effects of Somatostatin on Post-endoscopic Portal Hemodynamic in Cirrhotic Patients With Esophageal Gastric Varices
Brief Title: Effects of Somatostatin on Post-endoscopic Portal Hemodynamic in Cirrhotic Patients With Esophageal Gastric Varices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yunsheng Yang (Other)
Responsible Party: Sponsor-Investigator, Yunsheng Yang, chinese PLA General Hospital, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 0105467801
Record Dates: First submitted 2011-08-29; First posted 2011-08-31 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Esophageal Varices Secondary to Cirrhosis of Liver
MeSH Terms: interventions — Somatostatin; Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- endoscopic and somatostatin treatment (Experimental)
  Interventions: Drug: Somatostatin
- endoscopic therapy (Other)
  Interventions: Procedure: endoscopic therapy

INTERVENTIONS:
Drug: Somatostatin — giving stilamin 250ug/h after endoscopic therapy for 5 days
  Other Names: stilamin
  Arms: endoscopic and somatostatin treatment
Procedure: endoscopic therapy — gastroscope plus EIS/EVL/HI
  Other Names: antisterone,DHCT,albumin or antibiotics
  Arms: endoscopic therapy

SUMMARY:
The main complications of cirrhosis are ascites, esophageal varices and hepatic encephalopathy. About 30% to 70% patients with cirrhosis occur esophageal varices, and the most common complication is ascites. Somatostatin is used to treat esophageal for a long time, otherwise it could aslo prevent ascites. In the study, the investigators explore the effects of somatostatin on post-endoscopic portal hemodynamic in cirrhotic patients with esophageal gastric varices.

DETAILED DESCRIPTION:
126 patients will be enrolled in the study, 63 subjects will be randomized into the group A and the other will be into the group B.

Group A: endoscopic therapy and somatostatin treatment. Group B: endoscopic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis with esophageal gastric varices needed endoscopic therapy
* Age 18-75 years
* Informed written consent

Exclusion Criteria:

* Use of vasoactive drugs 24 hours before endoscopic treatment
* Use of B-blocker within 1 week
* Previous surgical or endoscopic treatment for esophageal gastric varices
* Hepatic encephalopathy,comatose status and any other disease which could not accept endoscopic therapy
* Gastro-renal vein shunt
* Severe hepatic hydrothorax
* Hepatocellular carcinoma with portal vein thrombosis
* Severe coagulation disorders
* Severe active bacteria infection
* Severe cardiovascular disease, including a history of acute myocardial infarction,heart block, heart failure
* Severe renal function insufficiency （Calculated Creatinine Clearance Rate (Ccr) <30ml/min）
* Severe co-morbidity that would affect short-term prognosis
* Pregnancy or lactation
* Allergy to any ingredient of trial medication
* Medical or psychological condition that would not permit the patient to complete the study or sign the informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Portal vein blood flow volume | change from baseline in portal vein blood flow volume after 7 days treatment
  Note:
  1. Portal vein blood flow volume will be measured by doppler ultrasound device.
  2. Values are the mean of three consecutive measurements.
  3. Frequency: PVF will be measured on baseline, day1, day 5 and day 7.
  4. All doppler studies will be carried out by a single experienced examiner who will be blinded to patient allocation.

SECONDARY OUTCOMES:
Portal vein diameter (PVD mm) | change from baseline in PDV after 7 days treatment
  Portal vein diameter will be measured by doppler ultrasound device.
Mean portal vein blood velocity (PVV cm/s) | change from baseline in PVV after 7 days treatment
  PVV will be measured by doppler ultrasound device.
Ascites volume | change from baseline after 7 days treatment
  Sonography detecting site: the middle point of the line between navel and the right side of anterior superior iliac spine(ASIS)

CONTACTS AND LOCATIONS:
Overall Officials: Yun Sh Yang, Pro., Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Site, Beijing, China